CLINICAL TRIAL: NCT04005131
Title: Effects of Upper Extremity Rehabilitation Robot and Transcranial Direct Current Stimulation on Upper Extremity Function Among Subjects With Chronic Stroke
Brief Title: Effects of Upper Extremity Rehabilitation Robot and Transcranial Direct Current Stimulation in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2018-01-003
Record Dates: First submitted 2019-06-18; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: stroke; transcranial direct current stimulation; upper extremity rehabilitation robot
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant does not know the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot and tDCS on-line (Experimental): Combined transcranial direct current stimulation(tDCS) on-line and upper extremity rehabilitation robot for 10 weeks
  Interventions: Device: Robot and tDCS on-line
- Robot and tDCS on-line after sham tDCS (Active Comparator): Combined sham tDCS and upper extremity rehabilitation robot for 5 weeks, followed by combined tDCS on-line and upper extremity rehabilitation robot for 5 weeks
  Interventions: Device: Robot and tDCS on-line after sham tDCS

INTERVENTIONS:
Device: Robot and tDCS on-line — Combined transcranial direct current stimulation(tDCS) on-line and upper extremity rehabilitation robot for 5 times a week for 10 weeks
  Arms: Robot and tDCS on-line
Device: Robot and tDCS on-line after sham tDCS — Combined sham tDCS and upper extremity rehabilitation robot for 5 times a week for 5 weeks, followed by combined tDCS on-line and upper extremity rehabilitation robot for 5 times a week for 5 weeks
  Arms: Robot and tDCS on-line after sham tDCS

SUMMARY:
Comparison of real transcranial direct current stimulation (tDCS) and sham tDCS combined with robot training for upper extremity rehabilitation in subjects with chronic stroke - delayed start study.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Onset ≥ 6 months
* Fugl-Meyer Assessment score ≥ 19
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* Severe upper extremity pain that could interfere with rehabilitation therapy
* Neurological disorders other than stroke that can cause motor deficits
* Uncontrolled severe medical conditions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
kinematic data during scale for the assessment | 5 weeks after baseline
  kinematic data during scale for the assessment and rating of ataxia using Trakstar (mean velocity, jerk, smoothness)

SECONDARY OUTCOMES:
kinematic data during scale for the assessment | baseline, 1 weeks after baseline, 5 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  kinematic data during scale for the assessment and rating of ataxia using Trakstar (mean velocity, jerk, smoothness)
Fugl-Meyer Assessment - upper extremity | baseline, 1 weeks after baseline, 5 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  indicator of the level of impairment of upper extremity, with higher scores indicating lower impairment
Wolf Motor Function Test | baseline, 1 weeks after baseline, 5 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  an activity indicator, has 15 items for testing functional ability
Motor activity log | baseline, 1 weeks after baseline, 5 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Assesses the use of the paretic arm and hand during activities of daily living in hemiparetic stroke patients.
Action reach arm test | baseline, 1 weeks after baseline, 5 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea